CLINICAL TRIAL: NCT04955834
Title: A Multicenter, Randomized, Open-label, Parallel-controlled Phase III Clinical Study to Compare the Efficacy and Safety of Insulin Degludec Injection Versus Tresiba® in Subjects With Type 2 Diabetes
Brief Title: A Clinical Study of Insulin Degludec Injection in Subjects With Type 2 Diabetes
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TQF2409-III-01
Record Dates: First submitted 2021-07-05; First posted 2021-07-09 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin degludec

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Insulin degludec injection (Experimental): Insulin degludec injection subcutaneous administration once daily for 26 weeks in combination with Oral antidiabetic drugs (OADs) used before.
  Interventions: Drug: Insulin degludec injection
- Tresiba® (Active Comparator): Insulin degludec injection（Tresiba®）subcutaneous administration once daily for 26 weeks in combination with Oral antidiabetic drugs (OADs) used before.
  Interventions: Drug: Tresiba®

INTERVENTIONS:
Drug: Insulin degludec injection — long-acting insulin
  Arms: Insulin degludec injection
Drug: Tresiba® — long-acting insulin
  Arms: Tresiba®

SUMMARY:
This study is a multi-center, randomized, open-label, parallel, positive-controlled registered clinical study,to evaluate the efficacy and safety of insulin degludec injection developed by Chia Tai Tianqing Pharmaceutical Group Co., Ltd.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes (diagnosed clinically) for at least 6 months.
2. Aged ≥18 and ≤70 years old, male or female.
3. Subjects who were treated with a stable dose of oral hypoglycemic agents for more than 3 months before the random visit.
4. HbA1c is in the range of 7.5% -11.0 % by local laboratory analysis.
5. Body mass index (BMI) ≥18 kg/m2 and ≤40kg/m2.
6. Patients must give informed consent to this study before the trial, and voluntarily sign an informed consent form.
7. Patients who can communicate well with the investigator and can complete the study in accordance with the research regulations.

Exclusion Criteria:

1. Diagnosed as type 1 diabetes or other types of diabetes.
2. Patients who have received insulin therapy for more than 7 days within 3 months before screening .
3. Patients who have received a thiazolidinedione (TZD) or GLP-1 receptor agonist within 3 months before screening.
4. Patients who are receiving or have received chronic (lasting more than 2 weeks) systemic glucocorticoid therapy (excluding topical drugs and inhaled preparations) within 3 months before the random visit.
5. Patients who are receiving or have received chronic (lasting more than 2 weeks) systemic glucocorticoid therapy (excluding topical drugs and inhaled preparations) within 3 months before the random visit.
6. Patients with hypoglycemia who have recurring severe events with conscious and/or physical changes within 3 months before screening and need help from others.
7. Those who have experienced acute metabolic complications (ketoacidosis, lactic acidosis, or hyperosmolar coma, etc.) within 3 months before screening.
8. Patients with obvious liver and kidney dysfunction.
9. Hemoglobin <100g/L.
10. When the virological test during the screening period shows that any of the following is met:

(1) HCV（hepatitis C virus） antibody is positive, and the HCV virus titer test value exceeds the upper limit of normal value; (2) HBsAg（Hepatitis B surface antigen） is positive and the HBV（hepatitis B virus） DNA test value exceeds the upper limit of normal; (3) HIV（human immunodeficiency virus） positive; (4) Active syphilis;

11. At the time of screening, there are thyroid diseases that have not been controlled with stable doses of drugs within 6 months, and the results of thyroid function tests during the screening period are abnormal and have clinical significance.

12. Uncontrolled or poorly treated high blood pressure.

13. Those with decompensated heart failure (NYHA class III and IV), unstable angina, stroke or transient ischemic attack, myocardial infarction, severe arrhythmia, cardiac surgery or blood vessel reconstruction (including coronary artery bypass grafting or percutaneous coronary intervention) occurred within 6 months before screening.

14. Those with proliferative retinopathy or macular degeneration (macular edema) that requires urgent treatment during screening.

15. Once diagnosed as malignant tumor (except for basal cell carcinoma or squamous cell skin cancer).

16. Patients with severe chronic gastrointestinal diseases (such as active peptic ulcer) and severe infections.

17. Those who are allergic to any ingredient in insulin deglu injection and Novota®.

18.Those who participated in any other clinical trials within 3 months before screening (excluding those who failed the screening or did not use study drugs for other reasons).

19. Pregnant women, lactating women, women of childbearing age who do not take appropriate contraceptive measures during the trial period (sterilization, intrauterine device, oral contraceptives or barrier contraception).

20. Those who are judged by the investigator to be unsuitable to participate in the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Estimated)
Dates: Start 2021-07-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change value of glycosylated hemoglobin (HbA1c) | Baseline and 26 weeks
  Change value of HbA1c from baseline following 26 weeks of therapy

SECONDARY OUTCOMES:
Percentage of patients achieving HbA1c ≤7% or HbA1c ≤6.5% | Baseline, week 26
  Percentage of patients in each arm achieving HbA1c ≤7% or HbA1c ≤6.5% after 26 weeks of treatment.
Change value of HbA1c | Baseline, week 14
  Change value of HbA1c from baseline following 14 weeks of therapy
Change value of fasting blood glucose | Baseline, week 14, week 26
  Change value of fasting blood glucose following 14 and 26 weeks of therapy
Adverse events (AEs) and serious adverse events (SAEs) | Baseline to week 26
  AEs and SAEs and their incidence during the 26-week treatment period, and then determine the correlation with the drug
Hypoglycemia | Baseline to week 26
  Frequency of severe or symptomatic hypoglycemia during the 26-week treatment period
Immunogenicity | Baseline, week 14, week 26
  The occurrence of immunogenicity during the 26-week treatment period by detecting Anti-Drug-Antibody(ADA).
Abnormal findings | Baseline to week 26
  Abnormal findings during the 26-week treatment period，including abnormal findings of blood routine test，blood biochemical test as well as other abnormal laboratory findings.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan